CLINICAL TRIAL: NCT04434586
Title: Contribution of Optical Coherence Tomography in the Endovascular Treatment of Femoral Occlusions
Acronym: TOCAF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018_88; 2019-A01055-52 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-06-08; First posted 2020-06-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Superficial Femoral Artery Stenosis; Claudication; Ischemic Leg
Keywords: femoral recanalization; optical coherence tomography (OCT); endovascular treatment; TASC-C,; TASC-D
MeSH Terms: conditions — Intermittent Claudication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- angiography 2D (Sham Comparator): Control group: an arteriography will be performed on the entire treated segment to assess the quality of the result, the application or not an active balloon will be left to the discretion of the operator. In case of application of the active balloon, a new arteriography before decision or not the use of stenting will be practiced. In case of stenting, an arteriographic final is performed.
  Interventions: Device: femoropopliteal revascularization for TASC C or TASC D lesion
- angiography 2D with OCT (Experimental): Experimental group: an arteriography and OCT acquisition on the entire treated segment to ensure the quality of the result, the application or not of an active ball will be left. In case of application of the active balloon, a new arteriography and OCT acquisition before decision or not the use of stenting will be practiced. In case of stenting, a final arteriography and then OCT acquisition are performed.
  Interventions: Device: femoropopliteal revascularization for TASC C or TASC D lesion

INTERVENTIONS:
Device: femoropopliteal revascularization for TASC C or TASC D lesion — Femoropopliteal revascularization: ATL or ATL/stenting for TASC C/D lesions. Control group: only angiography 2D final control. Experimental group: angiography + OCT control

SUMMARY:
This is a common care study. A study for evaluating the quality of balloon inflation and stent application will be performed in 2D angiography alone in the control group and then by 2D and OCT angiography for the experimental group. The benefit could be an improvement in the results of revascularization of femoropopliteal lesions thanks to OCT which allows a 3D visualization of the arterial lumen.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Femoral-popliteal lesion TASC-C or TASC-D de novo (F1 to P1)
* Starting lesion on the superficial femoral artery and not extending beyond the intercondylar notch (P2)
* ≥1 continuous permeable leg axis directly injecting the plantar arch
* Rutherford 2-5

Exclusion Criteria:

* Patient under personal protection regime (tutorship, guardianship)
* Absence of arterial axis in permeable leg
* Patient presenting a limb acute ischaemia (chart evolving since less than 14 days)
* Patient without favorable element to consider healing
* History of stents on the femoropopliteal axis
* History of femoropopliteal bypass
* Untreated stenosis ≥30% on the iliac axis and common femoral upstream
* Popliteal lesion beyond the intercondylar notch (P2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Primary patency rate at 1 year. | at 12 months (+/- 2months)
  The permeability rate is defined by the echodoppler criteria: PVS>2.4m/s or appearance of stenosis on the previously treated segment >70%.

SECONDARY OUTCOMES:
Primary patency rate at 1 year. | at 1month (+/- 10days), 6months (+/- 1month)
Target lesion revascularisation | at 1month (+/- 10days), 6months (+/- 1month) and 12 months (+/- 2months)
  corresponds to the occurrence of a re-intervention on the treated segment to maintain or restore permeability
Target vessel revascularisation | at 1month (+/- 10days), 6months (+/- 1month) and 12 months (+/- 2months)
  corresponds to the occurrence of a re-intervention on the previously treated artery, whatever the level, in order to maintain its permeability.
cost-effectiveness analyses | at 12 months (+/- 2months)
  Cost-effectiveness analysis between 2 therapeutic strategies: The costs related to each strategy are calculated taking into account the direct and indirect costs.

OTHER OUTCOMES:
Rutherford scale considered ordinal variable | at 1month (+/- 10days), 6months (+/- 1month) and 12 months (+/- 2months)
  Rutherford grade of 2-4 for their target leg. The Rutherford scale is an indicator for the severity of Peripheral Vascular Disease: 0 = no symptoms, 6 = functional foot is no longer salvageable (leading to foot amputation).
Variation in Ankle Brachial Index between randomization and 1, 6, 12 months on the revascularized limb in the study. | at 1month (+/- 10days), 6months (+/- 1month) and 12 months (+/- 2months)
  Ankle-brachial index defined as the ratio of the blood pressure at the ankle to the blood pressure in the upper arm
Variation in quality of life assessed by Walk Impairment Questionnary between randomization and 1, 6, 12 months. | at 1month (+/- 10days), 6months (+/- 1month) and 12 months (+/- 2months)
  a questionnaire for evaluating walking impairment in patients
  Parameters:
  * difficulty walking a distance during the past month
  * difficulty walking at a certain speed during the past month
  * symptoms associated with walking impairment
Variation in quality of life assessed by EQ5D scores between randomization and 1, 6, 12 months. | at 1month (+/- 10days), 6months (+/- 1month) and 12 months (+/- 2months)
  overall score on a numeric scale "check the box that best describes your health today", 5 themes (mobility, autonomy of the person, common activities, pain / discomfort, anxiety / depression)
Limb Rescue Rate | at 1month (+/- 10days), 6months (+/- 1month) and 12 months (+/- 2months)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Sobocinski, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Insitut Coeur-Poumon, CHU, Lille, France

REFERENCES:
- [Result] Dubosq M, Goueffic Y, Duhamel A, Denies F, Dervaux B, Goyault G, Sobocinski J. Optical Coherence Tomography Contribution Assessment in the Revascularization of Long Femoropopliteal Occlusive Lesions (TASC C and D): A Randomized Trial. Ann Vasc Surg. 2021 Jan;70:362-369. doi: 10.1016/j.avsg.2020.06.061. Epub 2020 Jul 4. PMID 32634565